CLINICAL TRIAL: NCT06093659
Title: A Randomised, Cross-Over, Nicotine Pharmacokinetic and Pharmacodynamic Study of Heated Tobacco and Heated Herbal Products Compared With Combustible Cigarettes
Brief Title: Nicotine Pharmacokinetic Study of Heated Tobacco and Heated Herbal Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial Brands PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NER 01/005
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Product use sequence ABECD (Experimental): Subjects use Product A on Day 1, Product B on Day 2, Product E on Day 3 and Product C on Day 4 and Product D on Day 5.
  Interventions: Other: Heated tobacco product with heated tobacco sticks (Product A); Other: Heated tobacco product with heated tobacco sticks (Product B); Other: Heated herbal product with nicotine-infused heated herbal sticks (Product C); Other: Heated herbal product with nicotine-infused heated herbal sticks (Product D); Other: Conventional Cigarette (Product E)
- Product use sequence BCADE (Experimental): Subjects use Product B on Day 1, Product C on Day 2, Product A on Day 3 and Product D on Day 4 and Product E on Day 5.
  Interventions: Other: Heated tobacco product with heated tobacco sticks (Product A); Other: Heated tobacco product with heated tobacco sticks (Product B); Other: Heated herbal product with nicotine-infused heated herbal sticks (Product C); Other: Heated herbal product with nicotine-infused heated herbal sticks (Product D); Other: Conventional Cigarette (Product E)
- Product use sequence CDBEA (Experimental): Subjects use Product C on Day 1, Product D on Day 2, Product B on Day 3 and Product E on Day 4 and Product A on Day 5.
  Interventions: Other: Heated tobacco product with heated tobacco sticks (Product A); Other: Heated tobacco product with heated tobacco sticks (Product B); Other: Heated herbal product with nicotine-infused heated herbal sticks (Product C); Other: Heated herbal product with nicotine-infused heated herbal sticks (Product D); Other: Conventional Cigarette (Product E)
- Product use sequence DECAB (Experimental): Subjects use Product D on Day 1, Product E on Day 2, Product C on Day 3 and Product A on Day 4 and Product B on Day 5.
  Interventions: Other: Heated tobacco product with heated tobacco sticks (Product A); Other: Heated tobacco product with heated tobacco sticks (Product B); Other: Heated herbal product with nicotine-infused heated herbal sticks (Product C); Other: Heated herbal product with nicotine-infused heated herbal sticks (Product D); Other: Conventional Cigarette (Product E)
- Product use sequence EADBC (Experimental): Subjects use Product E on Day 1, Product A on Day 2, Product D on Day 3 and Product B on Day 4 and Product C on Day 5.
  Interventions: Other: Heated tobacco product with heated tobacco sticks (Product A); Other: Heated tobacco product with heated tobacco sticks (Product B); Other: Heated herbal product with nicotine-infused heated herbal sticks (Product C); Other: Heated herbal product with nicotine-infused heated herbal sticks (Product D); Other: Conventional Cigarette (Product E)

INTERVENTIONS:
Other: Heated tobacco product with heated tobacco sticks (Product A) — Product A, used under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration), followed by an ad-libitum, 4-hour product use session on the same day.
Other: Heated tobacco product with heated tobacco sticks (Product B) — Product B, used under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration), followed by an ad-libitum, 4-hour product use session on the same day.
Other: Heated herbal product with nicotine-infused heated herbal sticks (Product C) — Product C, used under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration), followed by an ad-libitum, 4-hour product use session on the same day.
Other: Heated herbal product with nicotine-infused heated herbal sticks (Product D) — Product D, used under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration), followed by an ad-libitum, 4-hour product use session on the same day.
Other: Conventional Cigarette (Product E) — Subject's own brand combustible cigarette used under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration), followed by an ad-libitum, 4-hour product use session on the same day.

SUMMARY:
This is a randomised, cross-over, open-label, confinement study conducted in 25 adult male or female smokers of combustible cigarettes (CCs). The study investigates combustible cigarettes, heated tobacco products (HTPs), and Heated Herbal Products (HHPs), with endpoints including pharmacokinetic evaluation, and subjective effects.

Subjects will perform a Screening Visit and one Study Visit, including a 6-day confinement period.

ELIGIBILITY:
Inclusion Criteria:

* Reports smoking an average of at least 10 manufactured combustible (menthol or non-menthol) cigarettes per day for at least 12 months prior to Screening
* Has a positive urine cotinine (>500 ng/mL) at Screening
* Has an exhaled carbon monoxide >10 ppm at Screening
* Female subjects of childbearing potential must use contraception
* Male subjects must use contraception

Exclusion Criteria:

* Has a history or presence of clinically significant disease or condition that, in the opinion of the Investigator, would jeopardise the safety of the subject or impact the validity of the study results.
* Has a positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at Screening
* Has a body mass index (BMI) > 30.0 kg/m^2 or < 18.0 kg/m^2 at Screening
* Has a fever (>38.05°C) at Screening or check-in
* Has a history or presence of drug or alcohol abuse within 24 months of Check-in
* Pregnant or lactating females
* Has used any prescription smoking cessation treatments within 3 months prior to Check-in Is planning to quit smoking during the study or within the next 3 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Belfast, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Product Use Sequence ABECD: Subjects use Product A on Day 1, Product B on Day 2, Product E on Day 3 and Product C on Day 4 and Product D on Day 5. On each day, subjects completely use one single unit of the product (one stick, approximately 10 puffs, with 30-second interpuff intervals).
- Product Use Sequence BCADE: Subjects use Product B on Day 1, Product C on Day 2, Product A on Day 3 and Product D on Day 4 and Product E on Day 5. On each day, subjects completely use one single unit of the product (one stick, approximately 10 puffs, with 30-second interpuff intervals).
- Product Use Sequence CDBEA: Subjects use Product C on Day 1, Product D on Day 2, Product B on Day 3 and Product E on Day 4 and Product A on Day 5. On each day, subjects completely use one single unit of the product (one stick, approximately 10 puffs, with 30-second interpuff intervals).
- Product Use Sequence DECAB: Subjects use Product D on Day 1, Product E on Day 2, Product C on Day 3 and Product A on Day 4 and Product B on Day 5. On each day, subjects completely use one single unit of the product (one stick, approximately 10 puffs, with 30-second interpuff intervals).
- Product Use Sequence EADBC: Subjects use Product E on Day 1, Product A on Day 2, Product D on Day 3 and Product B on Day 4 and Product C on Day 5. On each day, subjects completely use one single unit of the product (one stick, approximately 10 puffs, with 30-second interpuff intervals).
Period: Overall Study
Arm/Group | Product Use Sequence ABECD | Product Use Sequence BCADE | Product Use Sequence CDBEA | Product Use Sequence DECAB | Product Use Sequence EADBC
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Product Use Sequence ABECD | Product Use Sequence BCADE | Product Use Sequence CDBEA | Product Use Sequence DECAB | Product Use Sequence EADBC | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (9.91) | 39.4 (8.62) | 43.2 (8.70) | 36.4 (12.58) | 37.8 (6.06) | 40.6 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 2 | 10
  Male | 3 | 3 | 3 | 3 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 5 | 5 | 5 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 5 | 5 | 5 | 5 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.46 (3.11) | 25.43 (1.57) | 25.63 (3.85) | 22.80 (2.72) | 26.15 (3.34) | 25.10 (3.00)

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Cmax
Description: Maximum measured plasma nicotine concentration, following the controlled product use session
Time Frame: 5 minutes pre-study product use and at 2, 4, 6, 8, 10, 15, 30, 45, 60, 120, and 240 minutes following the start of study product use
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Product A: All subjects after having used Product A under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
- Product B: All subjects after having used Product B under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
- Product C: All subjects after having used Product C under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
- Product D: All subjects after having used Product D under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
- Product E: All subjects after having used Product E under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
Arm/Group | Product A | Product B | Product C | Product D | Product E
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
ng/mL | 13.00 (9.80) | 12.97 (7.10) | 6.00 (3.28) | 6.87 (3.24) | 18.51 (10.05)

2. Primary Outcome: Nicotine AUCt
Description: The area under the concentration time curve for nicotine, from time 0 to the last observed non-zero concentration, following the controlled product use session
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*min/mL
Arm/Group | Product A | Product B | Product C | Product D | Product E
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
ng*min/mL | 716.3 (329.6) | 777.0 (289.4) | 363.9 (123.8) | 382.5 (145.0) | 1144.0 (427.9)

3. Secondary Outcome: Urge to Smoke Pre-use
Description: The subjects self-assess their urge to smoke by answering the question: "Right now, how much would you like to smoke a cigarette?" on a Visual Analog Scale (VAS), with scores of 0 to 100, with 0 being 'not at all' and 100 being 'a great deal'.
Time Frame: 10 minutes prior to the start of the product use session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Product A | Product B | Product C | Product D | Product E
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
units on a scale | 93.6 (10.7) | 94.0 (8.2) | 92.9 (8.8) | 91.9 (13.0) | 90.0 (17.8)

4. Secondary Outcome: Urge to Smoke Post-use
Description: as for outcome 3
Time Frame: At 240 minutes following the start of study product use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Product A | Product B | Product C | Product D | Product E
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
units on a scale | 91.4 (13.3) | 90.7 (11.9) | 88.7 (15.5) | 88.3 (18.6) | 87.6 (18.2)

5. Secondary Outcome: Urge to Smoke Emax
Description: The subjects self-assess their urge to smoke at defined time points by answering the question: "Right now, how much would you like to smoke a cigarette?" on a Visual Analog Scale (VAS), with scores of 0 to 100, with 0 being 'not at all' and 100 being 'A great deal'. Emax is calculated as the maximum absolute value of change from baseline (pre-use) (i.e., the maximum response) in VAS scores.
Time Frame: 10 minutes prior to the start of the product use session and at 2, 4, 6, 8, 10, 15, 30, 45, 60, 120, and 240 minutes following the start of study product use.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Product A | Product B | Product C | Product D | Product E
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
units on a scale | 56.0 (29.0) | 64.4 (29.0) | 43.0 (31.7) | 44.3 (28.9) | 69.2 (28.4)

6. Secondary Outcome: Puff Count
Description: Number of puffs taken during last 2 hours of the 4-hour ad-libitum product use session
Time Frame: Hours 2-4 of the 4-hour ad libitum product use session
Population: Topography parameters were only available for subsets of subjects due to technical issues with the puff topography analyser during the data recording process, which resulted in incomplete data capture for some participants.
Measure: Mean (Standard Deviation); unit: number of puffs
Groups:
- Product A: All subjects after having used Product A during last 2 hours of the 4-hour ad libitum product use session.
- Product B: All subjects after having used Product B during last 2 hours of the 4-hour ad libitum product use session.
- Product C: All subjects after having used Product C during last 2 hours of the 4-hour ad libitum product use session.
- Product D: All subjects after having used Product D during last 2 hours of the 4-hour ad libitum product use session.
- Product E: All subjects after having used Product E during last 2 hours of the 4-hour ad libitum product use session.
Arm/Group | Product A | Product B | Product C | Product D | Product E
Number analyzed (Participants) | 12 | 9 | 9 | 11 | 18
number of puffs | 30.3 (18.7) | 22.4 (14.3) | 32.4 (20.8) | 31.9 (13.7) | 20.2 (10.0)

ADVERSE EVENTS:
Time Frame: From Screening until follow-up visit 7 days after final product use (total of approx. 2 weeks)
Groups:
- Product A: All subjects having used Product A throughout the study.
- Product B: All subjects having used Product B throughout the study.
- Product C: All subjects having used Product C throughout the study.
- Product D: All subjects having used Product D throughout the study.
- Product E: All subjects having used Product E throughout the study.
Arm/Group | Product A | Product B | Product C | Product D | Product E
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 6/25 | 5/25 | 3/25 | 7/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Product A (N=25) | Product B (N=25) | Product C (N=25) | Product D (N=25) | Product E (N=25)
Nausea (Gastrointestinal disorders) | 4 | 0 | 1 | 2 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Catheter site irritation (General disorders) | 0 | 0 | 1 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Catheter site rash (General disorders) | 0 | 1 | 1 | 0 | 1
Catheter site swelling (General disorders) | 0 | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 2 | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT06093659/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT06093659/SAP_001.pdf